CLINICAL TRIAL: NCT07191314
Title: Long-term Evaluation of a Nasopharyngeal Airway
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Wallace H Coulter Center for Translational Research (Other)
Responsible Party: Principal Investigator, Louise O'Brien, Professor, Sleep Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00274782
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Sleep Apnea, Obstructive
Keywords: nasopharyngeal
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Nasopharyngeal airway device (Experimental): A nasopharyngeal airway obstructive sleep apnea ("NPA"-OSA) device will be used for two years at home.
  Interventions: Device: nasopharyngeal airway obstructive sleep apnea (NPA-OSA) device

INTERVENTIONS:
Device: nasopharyngeal airway obstructive sleep apnea (NPA-OSA) device — The NPA-OSA is a flexible, medical-grade silicone, tube-like device that is self-inserted into the user's nasopharyngeal airway through one nostril prior to sleep and worn throughout the night to reduce or alleviate snoring and obstructive sleep apnea.

SUMMARY:
This long-term follow-up study will permit continued device use for participants of the parent study (NCT06677151).

During study participation the study team will stay in contact with participants as necessary. Additionally, patients will undergo clinical follow-up as needed with their physician(s). At 12 months, participants will complete sleep questionnaires as part of this long-term follow-up period.

ELIGIBILITY:
Inclusion Criteria:

-Participants who completed the parent study (HUM00179497) and wish to continue using the NPA-OSA device.

Exclusion Criteria:

* The participants who were non-compliant with the NPA-OSA device during their participation in the parent study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in severity of apnea hypopnea index (AHI) | Baseline (day 0), 24 months
  The AHI is calculated by dividing the number of apnea events by the number of hours of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Louise M O'Brien, PhD, Principal Investigator — University of Michigan; David Zopf, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - Michigan Medicine, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No